CLINICAL TRIAL: NCT05841628
Title: Tolerability of 532 nm Laser Treatment of Port Wine Stains
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yakir Levin, MD, PhD, Instructor, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P003297
Record Dates: First submitted 2023-04-23; First posted 2023-05-03 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Port-Wine Stain
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Port wine stain (Experimental): The port wine stain will be treated with the DermaV laser. Within the single port wine stain, one area will be treated with standard settings (single pulse high fluence). Four other areas will be treated with multi-pulse low fluence settings. A sixth area will be an untreated control.
  Interventions: Device: 532 nm laser treatment

INTERVENTIONS:
Device: 532 nm laser treatment — The port wine birthmark will be treated with the DermaV 532 nm laser.

SUMMARY:
The goal of this study is to learn about treatment of port wine birthmarks treated with an FDA-approved 532 nm laser.

The main questions it aims to answer are:

* How well are the treatments tolerated?
* Are there differences in tolerability of the treatment when a single high fluence laser pulse is used (the standard treatment) versus using multiple low fluence pulses?
* Are there differences in results when using a single high fluence pulse versus multiple low fluence pulses?

type of study: Clinical Trial

Participants will undergo 3 monthly laser treatments with the 532 nm DermaV laser. Part of their birthmark will be treated with the standard single-pulse high fluence approach, and other parts will be treated with the multiple-pulse low fluence approach.

ELIGIBILITY:
Inclusion Criteria:

1. .Subject must be able to read, understand and sign the Informed Consent Form. 2. Female or Male, 18 to 75 years of age (inclusive). 3. Fitzpatrick Skin Type I - VI. 4. Have non-facial port wine stain covering at least 30cm2 area on the body. 5. Must be willing to have Lutronic DermaV treatments (532 nm) and able to adhere to the treatments, follow-up visit schedule, and post-treatment care instructions.

6. Willing to have very limited sun exposure and use sunscreen on the treatment area every day for the duration of the study, including the follow-up period.

7. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation (educational and/or marketing), publications, and any additional marketing purposes.

8. Agree to not undergo any other cosmetic procedure(s) or treatment(s) on the treated areas during the study and has no intention of having such procedures performed during the course of the study.

9. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.,

Exclusion Criteria:

1. Participation in a clinical trial of another drug, or device administered to the treatment area, within 3 months prior to enrollment or during the study.
2. Any type of prior cosmetic or port wine stain treatment to the target area within 3 months of study participation.
3. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including but not limited to, open lacerations or abrasions, hidradenitis, rash, infection , or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion).
4. Pregnant and/or breastfeeding, or planning to become pregnant.
5. Significant concurrent illness, such as diabetes mellitus, immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or using immunosuppressive medication.
6. Hypersensitivity to light exposure.
7. Any use of medication that is known to increase sensitivity to light according to the Investigator's discretion.
8. History of keloid scarring, hypertrophic scarring or abnormal wound healing or prone to bruising.
9. Has a history of squamous cell carcinoma or melanoma in the treatment area.
10. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders.
11. A history or active skin condition that in the opinion of the Investigator may interfere/confound with the treatment.
12. History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
13. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
14. History of pigmentary disorders, particularly tendency for hyper- or hypo- pigmentation, or any that are considered not acceptable by the study investigator.
15. Excessively tanned or active sun tan in area to be treated, or unable/unlikely to refrain from tanning during the study.
16. Excessive hair in the area to be treated (beards, sideburns, and/or moustache,) that would interfere with diagnosis, assessment, and treatment.
17. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study, including excessive alcohol or drug abuses, or a condition that would compromise the subject's ability to comply with the study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Degree of improvement | 6 months
  For each treatment area within the port wine stain, a blinded investigator will assess improvement (0 - 25%, 26 - 50%, 51 - 75%, 76 - 100%)

SECONDARY OUTCOMES:
Subject satisfaction | 6 months
  For each treatment area within the port wine stain, subject will assess satisfaction on a 1-4 scale
Side effects | 6 months
  subject and treating physician will assess side effects of treatment including pain, swelling, skin discoloration, scar

CONTACTS AND LOCATIONS:
Overall Officials: Yakir Levin, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Wellman Center for Photomedicine, Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared for this pilot study.